CLINICAL TRIAL: NCT03974425
Title: One Year Results of Switching to Aflibercept for Persistent Diabetic Macular Edema Resistant to Bevacizumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31184
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic macular edema resistant to Bevacizumab (Other): Patients resistant to 6 monthly Bevacizumab injection were switched to Aflibercept.
  Interventions: Drug: Aflibercept Injection [Eylea]

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — intravitreal injection of Aflibercept in resistant DME.

SUMMARY:
Purpose: The aim of this study is to evaluate the functional and anatomical effects of switching from Bevacizumab to Aflibercept in patients with persistent DME resistant to Bevacizumab.

Methods: Patients with DME refractory to Bevacizumab (1.25 mg/ 0.05 mL) were subsequently switched to Aflibercept (2.0 mg/0.05 ml). The included patients received 5 loading doses of intravitreal Aflibercept (2.0 mg/0.05 mL) (Eylea; Bayer, Berlin, Germany) given monthly. After the loading dose, Aflibercept was injected every 2 months. The follow up duration was one year.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients, older than 18years,
* center-involving DME, central macular thickness (CMT) >300 μm by spectral domain optical coherence tomography (SD-OCT) 1 month after the last Bevacizumab injection.
* The best corrected visual acuity must be better than 0.05 decimal visual acuity (1.3 log MAR). Only one eye from each patient was included in the study. If both eyes met the inclusion criteria, the eye with worse visual acuity was included.

Exclusion Criteria:

* Patients were excluded if they had dense media opacity, pregnancy, previous intravitreal steroid therapy.
* uncontrolled diabetes mellitus (HbA1c ≥ 10%) and prior intraocular surgery (with the exception of uneventful cataract surgery >6 months prior to conversion).
* Other exclusion criteria included active proliferative diabetic retinopathy, tractional maculopathy, macular ischemia and other ocular diseases: age-related macular degeneration, central/branch retinal vein occlusion, and glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
central macular thickness after one year | 12 months
  Optical Coherence Tomography changes after 12 months.

IPD SHARING:
Plan to Share IPD: No
protecting patient privacy